CLINICAL TRIAL: NCT05406661
Title: Registry of Local Recurrences After Breast-conserving Surgery in Portugal and Spain
Brief Title: Registry of Local Recurrences After Breast-conserving Surgery
Acronym: R_ReLoCC
Status: Not yet recruiting | Type: Observational
Sponsor: Universidade do Porto (Other)
Collaborators: Centro Hospitalar Universitário São João, EPE (Unknown)
Responsible Party: Sponsor
Other Study IDs: R_ReLoCC
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer Recurrent
Keywords: Breast cancer treatment; Local recurrences; Breast-conserving surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ReLoCC project is a prospective, multicenter, clinical study to register cases of local recurrence after breast-conserving surgery, in centers dedicated to the treatment of breast cancer, in Portugal and Spain.

The comparison of the results obtained will allow the optimization of the treatment, making it increasingly personalized.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients
2. Age > 18 years
3. Patients who have previously undergone breast-conserving surgery as part of the treatment of invasive or non-invasive (in situ) breast cancer

   1. and adjuvant breast RT: total (WBI) or partial (PBI)
   2. without adjuvant radiotherapy to the breast
4. Recent histological diagnosis of homolateral, invasive or non-invasive (in situ) breast carcinoma

Exclusion Criteria:

1. Male
2. Age < 18 years
3. Stage 4 at diagnosis
4. Patients operated outside the participating Centers and for whom it is not possible to obtain complete information regarding the primary treatment
5. History of other primary invasive malignant tumor (except non-melanoma skin carcinomas)
6. Patients already treated for another local recurrence of breast carcinoma
7. Absence of clinical follow-up and records in clinical process

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients
Study Population: Patients with local recurrence after breast-conserving surgery
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Determine prevalence of local recorrence of breast cancer after conserving surgery in Portugal and Spain | 2 years
  Number of cases per year
Follow-up of recurrences up to 5 years after treatment of first recurrence | 5 years
  Number of cases per year

SECONDARY OUTCOMES:
Identification of risk factors for local recurrence | On inclusion time (2 years)
  Frequency of risk factors
Identification of predictive and response factors | On inclusion time (2 years)
  Frequency of predictive factors
Determination of surgical morbidity of relapse treatment in follow up | From date of treatment until 30 days after treatment
  Identification of surgical morbidity
Assessment of patient quality of life | First and second year after treatment
  Validated questionnaire for quality of life by EORTC QLQ-C30-BR23

CONTACTS AND LOCATIONS:
Overall Officials: José Luis Fougo, MD, PhD, Study Director — Centro de Mama - Centro Hospitalar Universitário de São João

IPD SHARING:
Plan to Share IPD: No